CLINICAL TRIAL: NCT03672656
Title: Single Session of Pattern Scanning Laser Versus Multiple Sessions of Conventional Laser for Panretinal Photocoagulation in Diabetic Retinopathy: Efficacy, Safety and Painfulness
Brief Title: Pattern Laser Versus Conventional Laser in Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-OCNI-Pascal
Record Dates: First submitted 2018-09-07; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; patterns; low time of impulse; Pascal
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pattern scanning laser system Pascal (Experimental)
  Interventions: Device: lasercoagulation by Pascal system
- conventional laser (Active Comparator)
  Interventions: Device: conventional laser

INTERVENTIONS:
Device: lasercoagulation by Pascal system — pattern scanning laser system Pascal given in a single-session
  Arms: pattern scanning laser system Pascal
Device: conventional laser — conventional laser multiple-session treatment
  Arms: conventional laser

SUMMARY:
Purpose: To evaluate the clinical efficiency, safety and painfulness of retinal laser photocoagulation employing a pattern scanning laser system Pascal given in a single-session versus conventional laser multiple-session treatment of the same patient with diabetic retinopathy.

Methods: The cohort included 60 eyes in 30 patients treated at the Ophthalmology Clinic, Faculty Hospital Ostrava, from 2008 to 2013. Panretinal laser coagulation was performed on one eye using the multispot panretinal photocoagulation given in a single-session system Pascal (SSP) (OptiMedica, Santa Clara, California). On the other eye laser treatment was carried out by the classic conventional multiple-session method (MSM).

ELIGIBILITY:
Inclusion Criteria:

* Diabetic retinopathy

Exclusion Criteria:

* No

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2014-01-25 (Actual)

PRIMARY OUTCOMES:
Clinical efficiency - progression of diabetic retinopathy, scored by calculating of microaneurisms and intraretinal hemorrhages | 1 year
  progression of diabetic retinopathy after pattern PASCAL laser versus conventional laser. Each item is scored by calculating of microaneurisms and intraretinal hemorrhages
Pain assessed by NRS | 1 day
  painfulness of pattern PASCAL laser versus conventional laser Each item is scored 0-10 (0 - no pain, 10 - pain as bad as can be)

SECONDARY OUTCOMES:
Satisfaction assessed by the VAS | 1 day
  subjective satisfaction of the patient on dog 0 to 4 0 - not satisfied, 4 - very satisfied after pattern PASCAL laser versus conventional laser

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nemcansky J, Stepanov A, Nemcanska S, Masek P, Langrova H, Studnicka J. Single session of pattern scanning laser versus multiple sessions of conventional laser for panretinal photocoagulation in diabetic retinopathy: Efficacy, safety and painfulness. PLoS One. 2019 Jul 16;14(7):e0219282. doi: 10.1371/journal.pone.0219282. eCollection 2019. PMID 31310626